CLINICAL TRIAL: NCT06967012
Title: Efficacy and Safety of Zonisamide as a First Add-On Treatment in Focal Epileptic Seizures or Secondary Generalized Tonic-Clonic Seizures: A Clinical Study
Brief Title: A Clinical Study on the Efficacy and Safety of Zonisamide as a First Add-On Treatment in Epileptic Seizures
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-K171-02
Record Dates: First submitted 2025-02-02; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-11

CONDITIONS: Epilepsies, Partial; Epilepsy, Tonic-Clonic
Keywords: Zonisamide; Epilepsies, Partial; Epilepsy, Tonic-Clonic
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy, Tonic-Clonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Monotherapy and add-on therapy (Experimental): Zonisamide tablets are administered orally with the following dosage schedule: Weeks 1-2: 2 mg/kg/day, Weeks 3-4: 4 mg/kg/day, Weeks 5-6: 6 mg/kg/day. After the initial six weeks, the dosage is adjusted based on the patient's condition, with weekly increments of 1 mg/kg/day. The maintenance dose ranges from 4 to 6 mg/kg/day, administered in 1-2 divided doses daily. Participants weighing ≥50 kg receive adult-equivalent dosing.
  Interventions: Drug: Oral Zonisamide Therapy

INTERVENTIONS:
Drug: Oral Zonisamide Therapy — Zonisamide tablets are administered orally with the following dosage schedule: Weeks 1-2: 2 mg/kg/day, Weeks 3-4: 4 mg/kg/day, Weeks 5-6: 6 mg/kg/day. After the initial six weeks, the dosage is adjusted based on the patient's condition, with weekly increments of 1 mg/kg/day. The maintenance dose ranges from 4 to 6 mg/kg/day, administered in 1-2 divided doses daily. For children weighing ≥50 kg, the adult dosage should be used.

SUMMARY:
This study primarily aims to assess the efficacy and safety of zonisamide when used as an adjunctive therapy for focal epilepsy. The main questions it aims to answer are:

1. Does the frequency of epileptic seizures decrease after oral zonisamide， and does it improve cognitive function?
2. Are there any treatment-emergent adverse events associated with oral administration of zonisamide?

DETAILED DESCRIPTION:
This study primarily focuses on zonisamide, a drug originally developed as an antiepileptic and now used as an adjunctive treatment for focal epilepsy. Focal epilepsy is caused by abnormal electrical discharges in a specific area of the brain, which can lead to sudden loss of consciousness or muscle spasms. The main content of the study can be summarized as follows:

1. Research Purpose: To evaluate the efficacy and safety of zonisamide as an adjunctive treatment for focal epilepsy, especially for drug-resistant focal epilepsy.
2. Study Design: This is an open-label, observational study without a control group, planning to recruit 30 patients aged 1-14 years who have been stably taking one antiepileptic drug in the past 4 weeks but with poor results, and are now being considered for zonisamide treatment.
3. Treatment Plan: Patients will receive a gradually increasing dose of zonisamide, starting at 2 mg/kg/day and titrating up to 6 mg/kg/day, followed by a maintenance dose of 4-6 mg/kg/day depending on the patient's condition.
4. Effectiveness Evaluation: The efficacy of zonisamide is mainly assessed by comparing the change in seizure frequency before and after treatment and the proportion of patients whose seizure frequency is reduced by more than 50%.
5. Safety Assessment: The safety of zonisamide is assessed through physical examinations, weight monitoring, vital sign monitoring, and laboratory tests (including liver and kidney function and CBC).
6. Statistical Methods: Data analysis will be performed using SAS 9.4 statistical software, incorporating both descriptive and inferential statistics to assess the statistical significance of treatment effects.
7. Research Duration: August 1, 2024-July 31, 2027. This study is significant for exploring the potential of zonisamide as a new treatment plan, especially in combating epilepsy seizures that are difficult to control with traditional drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Consent to participate in the clinical trial, and the trial subject and/or legal guardian has signed the informed consent form.
2. Age 1-14 years, no gender restrictions.
3. Compliant with the diagnostic criteria for focal seizures and focal-to-bilateral tonic-clonic seizures as outlined by the International League Against Epilepsy (ILAE) in 2017.
4. Stable on one antiepileptic drug for ≥4 weeks, and deemed to be appropriate for the addition of zonisamide therapy by the investigator.
5. ≥ 2 episodes of generalized tonic-clonic seizures （secondary to focal epileptic seizures) per 28-day interval during the 8-week retrospective baseline period.

Exclusion Criteria:

1. History of zonisamide treatment.
2. History of allergy to sulfonamide drugs, zonisamide or any excipients.
3. History of drug/alcohol abuse.
4. History of suicide attempt or suicidal ideation within the past 6 months.
5. Current use of antidepressants, anxiolytics, or antipsychotics.
6. Diagnosed with progressive diseases affecting the brain and its functions.
7. Psychogenic non-epileptic seizures.
8. Diagnosed with severe pulmonary/hematologic diseases, malignant tumors, immunodeficiency, or psychiatric illnesses.
9. Have undergone epilepsy brain surgery or plan to undergo epilepsy surgery within the next 4 months.
10. Deemed to be unsuitable for participation in the trial by the investigator.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Primary Observational Indicators | Week 0±7day, Week 8±7day, Week 20±7day
  Change in seizure frequency: The reduction in seizure frequency over an average of four weeks during the maintenance period, compared with the retrospective baseline period, in patients with focal epilepsy with or without secondary generalized tonic-clonic seizures.
Primary Observational Indicators | Week 0±7day, Week 8±7day, Week 20±7day
  ≥50% response rate: The proportion of subjects achieving a ≥50% reduction in the average four-week seizure frequency during the maintenance period compared to the retrospective baseline period in patients with focal epilepsy with or without secondary generalized tonic-clonic seizures.

SECONDARY OUTCOMES:
Secondary Observational Indicators | Week 0±7day, Week 8±7day, Week 20±7day
  1. The percentage of patients achieving seizure-free status during the maintenance period in patients with focal epilepsy with or without secondary generalized tonic-clonic seizures.
  2. Retention rate: The percentage of patients who continue to take the medication within a specific time compared to the initial number of patients who started the medication.
Safety Evaluation | Week 0±7day, Week 8±7day, Week 20±7day
  Weight (kg)
Safety Evaluation | Week 0±7day, Week 8±7day, Week 20±7day
  blood pressure (mmHg)
Safety Evaluation | Week 0±7day, Week 8±7day, Week 20±7day
  Pulse (bpm)
Safety Evaluation | Week 0±7day, Week 8±7day, Week 20±7day
  Blood routine: WBC (/L), PLT (/L)
Safety Evaluation | Week 0±7day, Week 8±7day, Week 20±7day
  Liver function: ALT (U/L), AST (U/L), ALP (U/L)
Safety Evaluation | Week 0±7day, Week 8±7day, Week 20±7day
  Kidney function: Scr(μmol/L)
Safety Evaluation | Week 0±7day, Week 8±7day, Week 20±7day
  Blood routine: Hb (g/L)
Safety Evaluation | Week 0±7day, Week 8±7day, Week 20±7day
  Kidney function: UREA(mmol/L)
Safety Evaluation | Week 0±7day, Week 8±7day, Week 20±7day
  Liver function: TBIL (μmol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho D, Yu MS, Shin J, Lee J, Kim Y, Kang HC, Kim SH, Na D. A computational clinical decision-supporting system to suggest effective anti-epileptic drugs for pediatric epilepsy patients based on deep learning models using patient's medical history. BMC Med Inform Decis Mak. 2024 May 31;24(1):149. doi: 10.1186/s12911-024-02552-w. PMID 38822293